CLINICAL TRIAL: NCT02237742
Title: A Phase 1, Non-Randomized, Open-Label, Single-Dose, Single Period Study With Non-Pharmacologically Active Dose Of Pf-06427878 To Characterize Pharmacokinetics Following Intravenous Administration In Healthy, Adult, Male Subjects
Brief Title: A Study To Understand How The Body Reacts To A Low Dose Of PF-06427878 When Given In A Vein To Healthy, Adult, Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7871004; 2014-002626-12 (EudraCT Number)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-06427878 (Experimental)
  Interventions: Drug: PF-06427878

INTERVENTIONS:
Drug: PF-06427878 — Intravenous, 100 micrograms, single dose, 30 minute infusion

SUMMARY:
To determine how the body reacts to a low dose of PF-06427878 when given in a vein over 30 minutes to healthy, adult, males.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 18-55 years of age
2. BMI of 17.5-30.5 kg/m2

Exclusion Criteria:

1. History of drug or alcohol abuse within 2 years of screening
2. Subjects without suitable veins for multiple venipuncture/cannulation

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Day 1 Min 0,5,15,30,35,45,60,75,90, Hr 2,2.5,3.5,4.5,5.5,6.5,8.5,10.5,12.5,24.5
Area under the Plasma Concentration-Time Curve From Time Zero extrapolated to Infinite Time (AUCinf) | Day 1 Min 0,5,15,30,35,45,60,75,90, Hr 2,2.5,3.5,4.5,5.5,6.5,8.5,10.5,12.5,24.5
Maximum Observed Plasma Concentration (Cmax) | Day 1 Min 0,5,15,30,35,45,60,75,90, Hr 2,2.5,3.5,4.5,5.5,6.5,8.5,10.5,12.5,24.5
Plasma Terminal Elimination Half Life (t1/2) | Day 1 Min 0,5,15,30,35,45,60,75,90, Hr 2,2.5,3.5,4.5,5.5,6.5,8.5,10.5,12.5,24.5
Plasma Systemic Clearance (CL) | Day 1 Min 0,5,15,30,35,45,60,75,90, Hr 2,2.5,3.5,4.5,5.5,6.5,8.5,10.5,12.5,24.5
Plasma Volume of Distribution at Steady State (Vss) | Day 1 Min 0,5,15,30,35,45,60,75,90, Hr 2,2.5,3.5,4.5,5.5,6.5,8.5,10.5,12.5,24.5

SECONDARY OUTCOMES:
Amount of unchanged drug excreted in urine from time 0 to 12.5 hours (Ae12.5) | Day 1 Hr 0 to 12.5
Percent of dose excreted in urine as unchanged drug from time zero to 12.5 hours (Ae12.5%) | Day 1 Hr 0 to 12.5
Renal clearance (CLr) | Day 1 Hr 0 to 12.5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Quotient Clinical Ltd, Ruddington, Nottingham, United Kingdom